CLINICAL TRIAL: NCT05902767
Title: Nut Supplementation to Mitigate Post-stroke Cognitive Decline (NUT-me): a Pilot Study
Brief Title: Nut Supplementation to Mitigate Post-stroke Cognitive Decline
Acronym: NUT-me
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been extremely challenging.
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbara R. Cardoso, Senior Lecturer, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUT-me
Record Dates: First submitted 2023-05-18; First posted 2023-06-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Dementia
Keywords: dementia; cognitive decline; nuts
MeSH Terms: conditions — Stroke; Dementia; Cognitive Dysfunction | interventions — Nuts

STUDY DESIGN:
Intervention Model Description: The participants will be randomly assigned to one of the two study groups: Nuts of Control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nut Group (Experimental): Participants will receive a supply of mixed nuts containing: 1 Brazil nut (~3g), walnuts (15g), hazelnuts (7g), and almonds (7g) to be consumed daily for 90 days. They will also receive dietary counselling on how to follow the Australian Dietary Guidelines.
  Interventions: Other: Nuts
- Control Group (Other): Participants will follow the same protocol as the Nut group regarding appointments and collection of information. At the visits, they will receive dietary counselling on how to follow the Australian Dietary Guidelines
  Interventions: Other: Control

INTERVENTIONS:
Other: Nuts — * A mix of nuts containing 1 Brazil nut (~3g), walnuts (15g), hazelnuts (7g), and almonds (7g) to be consumed daily for 90 days.
  * Dietary counselling on how to follow the Australian Dietary Guidelines
  Arms: Nut Group
Other: Control — - Dietary counselling on how to follow the Australian Dietary Guidelines
  Arms: Control Group

SUMMARY:
Stroke is a strong risk factor for dementia, with up to 80% of individuals having lower cognitive function 5 years after a stroke event. However, having a stroke does not need to result in declining cognition if effective strategies to reduce the risk of post stroke dementia are identified. Diets containing nuts can reduce the risk of both dementia and stroke but have not been tested in stroke survivors. Therefore, this pilot study aims to determine whether eating nuts regularly reduces post-stroke cognitive decline and dementia. The NUT-me pilot study will supplement the diet of stroke survivors with a mix of nuts containing walnuts, hazelnuts, almonds and Brazil nuts for 3 months and assess the effects on cognition and health markers. The researchers predict that regular nut consumption will contribute to preserving post-stroke cognitive function in comparison to patients who do not consume nuts. The results of this novel pilot study will be used to guide a larger trial and provide a simple dietary strategy that stroke survivors can adopt to reduce post-stroke cognitive decline.

DETAILED DESCRIPTION:
This study will investigate the efficacy and feasibility of supplementing the habitual diet of stroke survivors with a supply of mixed nuts containing Brazil nut, walnuts, hazelnuts, and almonds to reduce post-stroke cognitive decline. The overall aim of this project will be achieved through the following objectives:

* Examine the feasibility through the assessment of compliance with the intervention and participants' perception of the study
* Investigate the efficacy of the intervention on cognitive decline, body composition and health outcomes (blood pressure, fasting glucose and insulin, and blood lipids) The investigators hypothesise that the inclusion of nuts is a simple dietary strategy that will slow post-stroke cognitive decline and that supplementation with nuts will improve body composition and health biomarkers of stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic stroke (first or recurrent stroke) in the last 6 months
* Able to attend 4 study visits over 3 months
* Motivation and willingness to participate in the study protocol
* No prior neurological or psychiatric disease, including dementia
* Can give informed consent and participate in cognitive testing

Exclusion Criteria:

* be < 18 years;
* have allergy to nuts
* have premorbid modified Rankin scale (mRS)≥4, denoting no severe disability
* incapable of giving consent
* have problems with mastication that preclude nut intake
* have habitual consumption of tree nuts (>2 servings/wk) in the previous 2 months
* have habitual consumption of alpha-linolenic acid supplements (fish oil, flaxseed oil, and/or soy lecithin)
* have dementia or psychiatric disease
* do not speak English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function Composite Score | 90 days
  Cognitive performance after the 90-day intervention will be assessed in comparison to baseline by using the NIH Toolbox Cognition Battery V3. This validated battery encompasses 15 tests that are combined to generate composite scores by age: Crystalised Composite (which includes picture vocabulary and oral reading recognition tests) and Fluid Composite (which includes dimensional change card sort, flanker, picture sequence memory, list sorting, and pattern comparison tests).The Cognitive Function Composite Score is a combination of both crystallized and fluid scores. Higher scores indicate better cognitive performance.

SECONDARY OUTCOMES:
Fluid Cognition Composite Score | 90 days
  Cognitive performance after the 90-day intervention will be assessed in comparison to baseline by using the NIH Toolbox Cognition Battery V3. This validated battery encompasses 15 tests that are combined to generate composite scores by age: Crystalised Composite (which includes picture vocabulary and oral reading recognition tests) and Fluid Composite (which includes dimensional change card sort, flanker, picture sequence memory, list sorting, and pattern comparison tests).The Cognitive Function Composite Score is a combination of both crystallized and fluid scores. Higher scores indicate better cognitive performance.
Crystallized Cognition Composite Score | 90 days
  Cognitive performance after the 90-day intervention will be assessed in comparison to baseline by using the NIH Toolbox Cognition Battery V3. This validated battery encompasses 15 tests that are combined to generate composite scores by age: Crystalised Composite (which includes picture vocabulary and oral reading recognition tests) and Fluid Composite (which includes dimensional change card sort, flanker, picture sequence memory, list sorting, and pattern comparison tests).The Cognitive Function Composite Score is a combination of both crystallized and fluid scores. Higher scores indicate better cognitive performance.
% body fat | 90 days
  Changes in % body fat measured using bioelectrical Impedance Analysis (BIA)
Depressive symptoms | 90 days
  Changes in the presence of depressive symptoms assessed by Patient Health Questionnaire (PHQ-9). The score ranges from zero to 27, with higher scores indicating worse depressive symptoms.
HOMA-IR | 90 days
  HOMA-IR is a measure of insulin resistance. It is calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Blood lipids | 90 days
  Changes in total cholesterol, LDL, HDL and triglycerides
Inflammatory markers | 90 days
  Changes in the composite of the following inflammatory markers: IL-6, IL-1β, IL-8, IL-10, and IL-1ra

CONTACTS AND LOCATIONS:
Overall Officials: Barbara R Cardoso, PhD, Principal Investigator — Department of Nutrition, Dietetics and Food - Monash University
Locations (1):
- Department of Nutrition, Dietetics and Food - Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and the generated data will be used only by the Principal Investigator as preliminary data in grant applications and potentially one publication (yet to be decided).